CLINICAL TRIAL: NCT04533217
Title: Palliative Treatment of Patients With Multiple Myeloma and Painful Vertebral Lesions. A Cross-sectoral Randomized Controlled Trial of Vertebroplasty in Addition to Regular Medical Treatment.
Brief Title: Examination of Vertebroplasty in Addition to Regular Treatment of Patients With Multiple Myeloma.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spine Centre of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: S-20200075
Record Dates: First submitted 2020-06-09; First posted 2020-08-31 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Vertebral Fracture; Multiple Myeloma
MeSH Terms: conditions — Spinal Fractures; Multiple Myeloma | interventions — Vertebroplasty

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vertebroplasty (Active Comparator): Patients treated with vertebroplasty in addition to regular medical treatment.
  Interventions: Procedure: Vertebroplasty
- Regular treatment (No Intervention): Patients treated with regular medical treatment.

INTERVENTIONS:
Procedure: Vertebroplasty — Injection of cement into vertebral lesion(s)
  Arms: Vertebroplasty

SUMMARY:
Patients with newly diagnosed or known multiple myeloma with newly diagnosed vertebral lesion(s) will be invited to participate in a cross-sectoral randomized controlled trial. The trial will compare two groups of patients which either receive regular medical treatment of their vertebral lesion(s) or vertebroplasty in addition to regular medical treatment. Our goal is to investigate the effectiveness of vertebroplasty and determine the role of surgical treatment in the overall treatment of patients with multiple myeloma and vertebral lesion(s).

DETAILED DESCRIPTION:
Patients identified by the attending consultant as eligible are invited to participate. Patients who express an interest in participating will be given written and oral information on the purpose, nature and implications of study-participation.

Possible candidates will be identified at the departments of Hematology where the patients are treated for their disease. All Danish departments of Hematology will be invited to participate.

The hematologist will inform the patient of the protocol and decide if they fulfil the inclusion and exclusion criteria. If the patient wishes to participate the hematologist will fill out screening forms regarding disease stage, lines of treatment, current disease status, bisphosphonate status, and pain relief treatment. The hematologist will refer the patient to their collaborating surgical department. The surgical department will decide if the patient has contraindications for surgery and inform the patient of the risk of the procedure.

If the patient decides to participate, he or she will fill out forms regarding ODI, VAS pain score, QoL.

Before randomization, the patients will be divided into two groups, stratifying between patients with known multiple myeloma with new diagnosed spine fracture and relevant pain ≤ 3 months prior to inclusion and patients with newly diagnosed multiple myeloma with new spine fracture.

Furthermore, to ensure balanced control and intervention groups the included patients at randomization will be stratified according to 1) panned PVP of 1 vs 2-4 levels, and 2) former vertebral fractures that are not planned treated with PVP.

The patients will be randomized to either PVP treatment or conservative treatment by drawing. It is therefore not possible for patients to choose between the treatments.

Patients randomized to vertebroplasty will be referred to a facility performing vertebroplasty. Patients randomized to non-vertebroplasty will receive the departments' usual care with the option to change treatment arm after 4 weeks.

The randomization will be performed by the diagnosing clinician, but orchestrated by one individual central to the clinics. The clinics will receive sealed envelopes containing the choice of randomization equally divided between PVP and conservative treatment. When all sealed envelopes have been used for randomization, the clinics will receive new envelopes.

It will not be possible to randomize more than one patient at a time. All patients will be contacted by a research nurse on a weekly basis the first 12 weeks after enrolment and after 3 and 12 months.

All patients randomized to vertebroplasty will undergo standard operative treatment involving a standard scheduled outpatient clinical control with the surgeon 12-weeks post-operative including long-standing radiographs of the spine.

ELIGIBILITY:
Inclusion Criteria:

* known multiple myeloma
* verified lesion(s) between Th6-L5
* 4 or less fractures
* relevant pain in 3 months or less
* vertebroplasty can be performed in one procedure
* VAS 5 or more

Exclusion Criteria:

* presence of neurologic deficit
* psychological or psychiatric disorder hat is expected to interfere with compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in back-specific disability | 4 weeks post-initiation of treatment
  Oswestry Disability Index v2.1 (ODI): Each section is scored on a 0-5 scale, with 5 representing the highest disability.

SECONDARY OUTCOMES:
Improvement in back-specific disability | Up to 12 months post-initiation of treatment
  ODI
Back and leg pain | Up to 12 months post-initiation of treatment
  Visual Analogue Scale (VAS): 0-100 scale, with 100 representing the largest amount of pain
Movement, personal care, usual activities, pain/discomfort, depression/anxiety | Up to 12 months post-initiation of treatment
  Self-reported questionnaire on quality of life using:
  - European Quality of Life - 5 Dimension (EQ-5D): 0-2 scale, with 2 representing the highest disability
  EQ-5D contains questions on topics contributing to the overall feeling of quality of life:
  * movement
  * personal care
  * usual activities (ex. occupation, family activities)
  * pain/discomfort
  * depression/anxiety.
Long-term stability of treated vertebra(e) | 12 months post-initiation of treatment
  X-rays will be used to analyze long-term stability.
General health services | Up to 12 moths post-initiation of treatment
  General questionnaires on wether or not and to what extend the patients have been using general health services.

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel Andersen, Professor, Principal Investigator — Centre of Spine Surgery and Research, Middelfart Hospital
Locations (1):
- Center for Spine Surgery and Research, Middelfart, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All data of long-term value will be stored, e.g. for use in future studies on shorter-term or long-term follow-up or reuse.
  Metadata and anonymized data will be available for other researchers if possible due to confidentiality and GDPR.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Wickstroem LA, Carreon L, Lund T, Abildgaard N, Lorenzen MD, Andersen MO. Vertebroplasty in patients with multiple myeloma with vertebral compression fractures: protocol for a single-blind randomised controlled trial. BMJ Open. 2021 Sep 6;11(9):e045854. doi: 10.1136/bmjopen-2020-045854. PMID 34489267

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-13): https://cdn.clinicaltrials.gov/large-docs/17/NCT04533217/Prot_SAP_000.pdf